CLINICAL TRIAL: NCT02463188
Title: Promoting Sleep to Prevent Substance Use in Adolescence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5R34DA035349-02 (NIH)
Record Dates: First submitted 2015-05-26; First posted 2015-06-04 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Sleep; Substance Use
Keywords: Sleep; Substance Use; Adolescents
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep Fitness Intervention (Experimental): The intervention consists of 5-7 sessions on sleep science, the connection between sleep and substance use, behavior change strategies, and motivation to change behavior.
  Interventions: Behavioral: Sleep Fitness Intervention
- Psychoeducation (PE) (No Intervention): The control classes will receive an 1-session psycho-educational (PE) intervention that provides information on sleep but does not provide guidance for implementing behavior change and does not explicitly teach about sleep's relationship to substance use.

INTERVENTIONS:
Behavioral: Sleep Fitness Intervention — The intervention consists of 5-7 sessions. Each session includes interactive and small group discussions. The intervention also includes lessons on sleep science, behavior change strategies, and one-on-one motivational interviews on behavior change motivation.
  Arms: Sleep Fitness Intervention

SUMMARY:
The goal is to adapt and refine an innovative, developmentally-appropriate universal health promotion intervention to reduce insufficient sleep among adolescents aged 14 to 16, while engaging teens in the adaptation process to maximize the relevance, appeal, and effectiveness of the program for diverse school settings.

DETAILED DESCRIPTION:
The goal is to adapt and refine an innovative, developmentally-appropriate universal health promotion intervention to reduce insufficient sleep among adolescents aged 14 to 16, while engaging teens in the adaptation process to maximize the relevance, appeal, and effectiveness of the program for diverse school settings.

The investigators aim to conduct a pilot feasibility randomized controlled trial (RCT) among adolescents (n = 300) who will be randomized to Sleep Fitness (SF) or Sleep Education (SE) to obtain effect size estimates in preparation for a larger scale intervention study. This pilot trial is designed to obtain preliminary data for the following hypotheses:

SF, compared to SE, will produce greater pre-post improvement in sleep after treatment and at 6 month follow-up (with the possibility of a 12 month follow-up for a subset of participants, depending on resources).

SF, compared to SE, will produce greater pre-post reductions in substance use after treatment and at 6 month follow-up (with the possibility of a 12 month follow-up for a subset of participants, depending on resources).

SF, compared to SE, will produce greater pre-post improvement on selected mental health outcomes (anxiety, depression) after treatment and at 6 month follow-up (with the possibility of a 12 month follow-up for a subset of participants, depending on resources).

ELIGIBILITY:
Inclusion and exclusion criteria are considered at the level of schools, classes, and students.

Inclusion Criteria:

* Schools: Only general education high schools, not "newcomer" schools that target immigrants with limited English ability. Our rationale is that we need students to read and understand English well enough to complete our study measures and understand the intervention.
* Classes: After the selection of schools, we will select classes that are representative of the school, insofar as they do not reflect Advanced Placement or remedial classes and utilize similar criteria for admission to the classes (e.g. health, advisory) so that we minimize differences between the classes in the study.
* Students: All participants must receive parental consent, provide their own consent, and must have sufficient English language ability

Exclusion Criteria:

* We propose no exclusion criteria for students who receive parental consent, provide their own assent, and have sufficient English language ability.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2014-02; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Primary Sleep | Change from baseline to post-intervention, which will be conducted between 5 and 8 weeks after the baseline assessment, and at 6 month follow-up (with the possibility of a 12 month follow-up for a subset of participants, depending on resources)
  Sleep Diary 1 Week: Total sleep time (Average of weeknights)
Primary Substance Use | Change from baseline to post-intervention, which will be conducted between 5 and 8 weeks after the baseline assessment, and at 6 month follow-up (with the possibility of a 12 month follow-up for a subset of participants, depending on resources)
  Measures from Monitoring the Future: 30-day use

SECONDARY OUTCOMES:
Depressive Symptoms | Change from baseline to post-intervention, which will be conducted between 5 and 8 weeks after the baseline assessment, and at 6 month follow-up (with the possibility of a 12 month follow-up for a subset of participants, depending on resources)
  Center for Epidemiologic Studies- Depression
Anxiety Symptoms | Change from baseline to post-intervention, which will be conducted between 5 and 8 weeks after the baseline assessment, and at 6 month follow-up (with the possibility of a 12 month follow-up for a subset of participants, depending on resources)
  Revised Children's Manifest Anxiety Scale

OTHER OUTCOMES:
Sleep | Change from baseline to post-intervention, which will be conducted between 5 and 8 weeks after the baseline assessment, and at 6 month follow-up (with the possibility of a 12 month follow-up for a subset of participants, depending on resources)
  Sleep Diary 1 Week: Total sleep time (average of weekend nights); Difference between average TST on weeknights and average TST on weekend nights; Average weeknight bedtime; Average weekend bedtime, Difference between average weeknight bedtime and average weekend bedtime; Average weekend rise time; Difference between average weekday rise time and average weekend rise time; Sleep Onset Latency (calculated separately for weeknights and weekend nights) and Wake After Sleep Onset (calculated separately for weeknights and weekend nights) to create Total Wake Time for weeknights, weekends and to also compute the discrepancy between weeknights and weekend nights; Sleep efficiency.
  Pittsburgh Sleep Quality Index: Total Score and subscale scores.
Substance Use | Change from baseline to post-intervention, which will be conducted between 5 and 8 weeks after the baseline assessment, and at 6 month follow-up (with the possibility of a 12 month follow-up for a subset of participants, depending on resources)
  Measures from Monitoring the Future: Substance use at all other applicable time points (in last day, in last week, in last 12 months, in lifetime).
Sleep Motivation (moderator) | Change from baseline to post-intervention, which will be conducted between 5 and 8 weeks after the baseline assessment, and at 6 month follow-up (with the possibility of a 12 month follow-up for a subset of participants, depending on resources)
  Measure developed for this study to assess motivation to change sleep behaviors.
Sleep Self-Efficacy (moderator) | Change from baseline to post-intervention, which will be conducted between 5 and 8 weeks after the baseline assessment, and at 6 month follow-up (with the possibility of a 12 month follow-up for a subset of participants, depending on resources)
  Measure developed for this study to assess self-efficacy to change sleep behaviors.
Perceived Stress (moderator) | Change from baseline to post-intervention, which will be conducted between 5 and 8 weeks after the baseline assessment, and at 6 month follow-up (with the possibility of a 12 month follow-up for a subset of participants, depending on resources)
  Daily Hassles Scale: Total score
Peer Norms of Substance Use (moderator) | Change from baseline to post-intervention, which will be conducted between 5 and 8 weeks after the baseline assessment, and at 6 month follow-up (with the possibility of a 12 month follow-up for a subset of participants, depending on resources)
  Monitoring the Future: Norms and Availability of Substance Use

CONTACTS AND LOCATIONS:
Overall Officials: Allison Harvey, PhD, Principal Investigator — University of California, Berkeley; Emily Ozer, PhD, Principal Investigator — University of California, Berkeley
Locations (1):
- University of California at Berkeley, Berkeley, California, United States